CLINICAL TRIAL: NCT04909957
Title: Prediction of Lymph Node Invasion in Patients Operated on for Prostate Adenocarcinoma
Brief Title: Prediction of Lymph Node Invasion for Prostate Adenocarcinoma
Acronym: PRED-NCHIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0290
Record Dates: First submitted 2021-01-26; First posted 2021-06-02 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: MRI; Lymph node

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Absence of invaded lymph node after extensive lymph node dissection: Absence of invaded lymph node after extensive lymph node dissection
- Presence of invaded lymph node after extensive lymph node dissection: Presence of invaded lymph node after extensive lymph node dissection

SUMMARY:
Despite lymph node involvement (LNI) being one of the main prognostic factors in patients with prostate cancer (PCa), pelvic lymph node irradiation remains debated, possibly due to an insufficient selection of patients. Significant advances in LNI risk modelling have been achieved with the addition of visual interpretation of magnetic resonance imaging (MRI) data, but it is likely that quantitative analysis could further improve prediction models. In this study, the investigators aimed to develop and internally validate a novel LNI risk prediction model based on radiomic features extracted from pre-operative multimodal MRI.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate treated by prostatectomy with extensive lymph node dissection
* Available pre-operative +/- PET choline

Exclusion Criteria:

* Unanalyzable pre-operative MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of patients operated on for an adenocarcinoma of the prostate by radical prostatectomy with extensive lymph node dissection and for whom pre-operative MRI is available and analyzable.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Predicted risk of lymph-node involvement vs Briganti 2017 | immediately after the intervention/procedure/surgery
  Comparison between the predicted risk of lymph node involvement based on the new algorithm and the predicted risk with the Briganti 2017

SECONDARY OUTCOMES:
Predicted risk of lymph-node involvement vs Briganti 2012, Briganti 2018, Briganti 2019 and MSKCC | immediately after the intervention/procedure/surgery
  Comparison between the predicted risk of lymph node involvement based on the new algorithm and the predicted risk with the Briganti 2012, Briganti 2018, Briganti 2019 and MSKCC
Biochemical recurrence free survival | immediately after the intervention/procedure/surgery
  Prediction of Biochemical recurrence free survival
Extra-prostatic disease | immediately after the intervention/procedure/surgery
  Prediction of Extra-prostatic disease
Seminal vesicle invasion | immediately after the intervention/procedure/surgery
  Prediction of Seminal vesicle invasion
Automatic segmentation of the index lesion | immediately after the intervention/procedure/surgery
  Comparison between a manual segmentation of the index lesion and an automatic segmentation

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three month and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.